CLINICAL TRIAL: NCT07076706
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of CG2001 in Chinese Adult Male Participants With Androgenetic Alopecia
Brief Title: Clinical Trial to Evaluate CG2001 in Chinese Adult Male Participants With Androgenetic Alopecia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Dayspring Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG2001-C-2
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Male Pattern of Hair Loss, Androgenic Alopecia; Androgenetic Alopecia (AGA)
Keywords: minoxidil; finasteride
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Minoxidil and low dose finasteride or placebo (Experimental): CG2001(5%minoxidil+0.075%finasteride) or placebo twice daily
  Interventions: Drug: minoxidil + finasteride; Drug: Placebo foam
- Minoxidil and high dose finasteride or placebo (Experimental): CG2001(5%minoxidil+0.1%finasteride) or placebo twice daily
  Interventions: Drug: minoxidil + finasteride; Drug: Placebo foam
- Minoxidil and low dose finasteride (Experimental): CG2001(5%minoxidil+0..075%finasteride) twice daily
  Interventions: Drug: minoxidil + finasteride
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo foam

INTERVENTIONS:
Drug: minoxidil + finasteride — topical foam: 5%minoxidil+0.075%finasteride
  Arms: Minoxidil and low dose finasteride; Minoxidil and low dose finasteride or placebo
Drug: minoxidil + finasteride — topical foam: 5%minoxidil+0.1%finasteride
  Arms: Minoxidil and high dose finasteride or placebo
Drug: Placebo foam — Topical placebo foam
  Arms: Minoxidil and high dose finasteride or placebo; Minoxidil and low dose finasteride or placebo; Placebo

SUMMARY:
The main objectives of this study are to preliminarily evaluate the effectiveness of CG2001 in treating Chinese adult male AGA participants, determine the recommended dose for Phase III clinical studies, and evaluate the safety of CG2001 at the target dose.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria can be included in this study:

1. Voluntarily sign the Informed Consent Form (ICF) approved by the Ethics Committee (IEC) before any study procedures begin. Participant who can understand and comply with the requirements of the protocol and agree to participate in all study visits;
2. Male participant, aged 18 to 65 years (including the critical value) when signing the ICF;
3. Participant diagnosed with androgenic alopecia, manifested as frontal hairline recession or hair loss in the vertex scalp area, corresponding to the Hamilton-Norwood classification diagnosis of grade III vertex type (i.e. grade IIIv), grade IV and grade V;
4. Willing and able to complete all study assessments and comply with the protocol study schedule and restrictions, such as the participant is willing to shave the target evaluation area during the study, be marked by the researcher and maintain the same hair color;
5. Participant agrees to use appropriate medical contraceptive methods to avoid pregnancy in female partners from the signing of the ICF until 28 days after the last dose.

Exclusion Criteria:

Before screening or administration, participants who meet any of the following criteria will not be included in this study:

1. Allergic to any component of minoxidil, finasteride or excipients (such as a history of alcohol allergy), or allergic constitution;
2. According to the researcher's judgment, the participant's head has any of the following conditions that may interfere with the study evaluation:

   A. History of scalp skin abnormalities or scalp skin diseases, such as obvious dermatitis, trauma or infection near the administration site; B. White hair in the hair loss area that obviously interferes with the study evaluation; C. Secondary hair loss, such as hair loss caused by malnutrition, drugs, endocrine (hypothyroidism or hyperthyroidism, parathyroid or pituitary dysfunction), iron deficiency anemia and systemic lupus erythematosus; D. Hair loss caused by other reasons other than androgenic alopecia, such as alopecia areata, scarring alopecia, trichotillomania, telogen effluvium, or sudden increase in hair loss within 3 months before screening;
3. Regarding the history of previous treatment, any of the following conditions may interfere with the study evaluation:

   A. Use of oral finasteride, dutasteride or similar products for androgenic alopecia within 1 year before screening; B. Use of topical minoxidil, local scalp radiation, phototherapy/laser or local injection of autologous platelet-rich plasma (PRP) within 6 months before screening; C. Underwent general anesthesia within 3 months before screening; D. Use of systemic or topical scalp corticosteroids or synthetic steroids, or other drugs that affect androgenic alopecia within 4 weeks before screening or within 5 half-lives of the drug used (whichever is longer); E. Use of medical shampoos or solutions containing other ingredients such as ketoconazole or similar ingredients that may interfere with efficacy evaluation within 1 week before the first medication; F. Participants who have had hair transplantation, hair extensions or hair weaving before screening; or plan to have hair transplantation, hair extensions or hair weaving during the study treatment; or need to wear a wig for a long time; G. Participants who plan to use treatments related to hair growth and may affect prolactin levels; H. Participants who have used minoxidil regularly for ≥4 months but have not been effective; I. Participants who have received CG2001 treatment before.
4. Other diseases with poorly controlled conditions that may affect the safety and efficacy evaluation of the trial drugs, such as malignant tumors, or poorly controlled diseases in the circulatory system, nervous system, blood system, digestive system (such as inflammatory bowel disease), immune system, mental system, etc. (except for completely resected carcinoma in situ, localized prostate cancer that has received radical treatment and has no disease recurrence, completely resected basal cell or squamous cell skin cancer, malignant melanoma with a complete remission time of more than 10 years, and other malignant tumors with a complete remission time of more than 5 years); or participants who plan to undergo surgery during the study; or within 3 months before screening, the weight loss exceeds 10% of their original body weight;
5. Physical examination, vital signs, 12-lead electrocardiogram (ECG), blood routine, urine routine, blood biochemistry, and sex hormone test results during the screening period are abnormal and clinically significant (especially for participants with anemia), and the researchers judge that it will affect the safety assessment;
6. History of drug abuse, alcoholism or drug abuse within 5 years before screening (Note: alcoholism includes binge drinking and heavy drinking. Binge drinking means that men drink 5 or more alcoholic drinks in about 2 hours at a time; heavy drinking or harmful drinking means that men drink 4 or more alcoholic drinks on any day, or the average daily alcohol intake of male drinkers is ≥61g; "cup" here means "standard cup", that is, 1 standard cup equals 10 grams of pure alcohol, 1 bottle of 750 ml wine is equivalent to 9 standard cups, 1 bottle of beer is equivalent to 2 standard cups, 1 bottle of 500 ml yellow wine (rice wine) is equivalent to 6 standard cups, 1 liang of 52-degree liquor is equivalent to 2 standard cups, 1 liang of 45-degree liquor is equivalent to 1.8 standard cups, 1 liang of 38-degree liquor is equivalent to 1.5 standard cups, and the number of grams of alcohol intake is equal to the number of milliliters of alcohol consumed × alcohol content × 0.8);
7. Participated in or is participating in other interventional clinical trials (including drugs and medical devices) within 1 month before screening;
8. The researcher believes that there are any other reasons that make the participants unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the non-vellus target area hair count(TAHC) at 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Hair Growth Questionnaire | 6, 12, 18, 24 weeks
  Questionnaire assessing hair condition by participant. The score ranges from 7 to 38, higher scores mean a worse outcome.
Participant self assessment of treatment satisfaction | 6, ,12, 18, 24 weeks
  Treatment satisfaction will be measured with the "Patient Treatment-Effect Satisfaction Evaluation Form", a single-item, self-administered questionnaire with the score ranges from -3 to +3, where a higher score mean a highr satisfaction.
Investigator Global Assessment(IGA) | 6, 12, 18, 24 weeks
  Assessment made by investigator about the global condition of participant's hair. The value ranges from 0 to 4, higher score means a worse outcome.
Change from baseline in non-vellus target area hair count(TAHC) | 6, 12, 18 weeks
Change from baseline in Target Area Hair Width(TAHW) | 6, 12, 18, 24 weeks
  Target Area Hair Width (TAHW) is the cumulative hair diameter per unit area in the target area
Change from baseline in terminal-vellus ratio | 6, 12, 18, 24 weeks
Adverse events | up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, MD, PhD, Study Chair — Peking University People's Hospital; Cheng Zhou, MD, PhD, Study Chair — Peking University People's Hospital
Locations (8):
- China (8):
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangxi Provincial Dermatology Hospital, Nanchang, Jiangxi
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Peking University People's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No